CLINICAL TRIAL: NCT00180518
Title: Prospective, Non-Randomized, Multi-Center, Single-Arm Trial to Assess Safety & Efficacy of the Acculink Carotid Stent System With the Accunet Embolic Protection System in High-Risk Patients With Carotid Artery Lesions.
Brief Title: ACCULINK for Revascularization of Carotids in High Risk Patients "The ARCHeR Trial"
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Abbott Vascular, Abbott Vascular
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 99-706
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2008-09-12 (Estimated); Status verified 2008-09

CONDITIONS: Carotid Atherosclerosis; Carotid Artery Disease
Keywords: Carotid artery disease; High risk; High surgical risk
MeSH Terms: conditions — Carotid Artery Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): To evaluate the safety and efficacy of the over-the-wire (OTW) ACCULINK (tm) System in patients deemed to be either at high risk or unsuitable for carotid endarterectomy (CEA) To evaluate the efficacy of the OTW ACCUNET System in patients deemed to be either at high risk or unsuitable for carotid endarterectomy (CEA).
  To demonstrate equivalence in the safety and performance of the RX ACCULINK Carotid Stent System and RX ACCUNET Embolic Protection System and the corresponding OTW devices.
  Interventions: Device: Over-the-wire & Rapid Exchange ACCULINK (tm) Carotid Stent & ACCUNET (tm) embolic protection system

INTERVENTIONS:
Device: Over-the-wire & Rapid Exchange ACCULINK (tm) Carotid Stent & ACCUNET (tm) embolic protection system — Two rapid exchange devices will be evaluated: the RX ACCUNET Embolic Protection System ("RX ACCUNET") and the RX ACCULINK Carotid Stent System ("RX ACCULINK").
  The RX ACCUNET Embolic Protection System is intended to facilitate the placement of diagnostic and therapeutic devices during interventional procedures and to capture embolic material that may be present during carotid artery interventional procedures.
  The RX ACCULINK™ Carotid Stent System is intended for the treatment of carotid artery stenosis in the internal carotid artery (ICA), with or without involvement of the contiguous common carotid artery (CCA), in asymptomatic patients and symptomatic patients.

SUMMARY:
1. To evaluate the safety and efficacy of the over-the-wire (OTW) ACCULINK (tm) System in patients deemed to be either at high risk or unsuitable for carotid endarterectomy (CEA)
2. To evaluate the efficacy of the OTW ACCUNET System in patients deemed to be either at high risk or unsuitable for carotid endarterectomy (CEA).
3. To demonstrate equivalence in the safety and performance of the RX ACCULINK Carotid Stent System and RX ACCUNET Embolic Protection System and the corresponding OTW devices.

DETAILED DESCRIPTION:
The purpose of the study is to demonstrate equivalence in the safety and performance of the RX ACCUNET when used with the RX ACCULINK, to that of the ACCULINK and ACCUNET devices, in the treatment of high risk surgical patients and patients with anatomical risks who require treatment for carotid artery disease.

Patients in ARCHeR RX will be followed after the index procedure at one, six and 12 months. Equivalence in safety will be demonstrated by comparing 30-day rates of DSMI for ARCHeR Amendment 2 and ARCHeR RX. Secondary analyses will be performed on the rate of ipsilateral stroke between 31 days and 12 months, target lesion revascularization at six and 12 months, acute device success for the RX ACCULINK and RX ACCUNET Systems, clinical success, and access site complications requiring treatment. Additionally, the stented segment will be evaluated by carotid duplex ultrasound at six and 12 months. Serious adverse events (SAE) of death or ipsilateral stroke that occur anytime during the follow-up period will be identified and reported, and will be adjudicated if indicated.

ELIGIBILITY:
Inclusion Criteria:

1. Patient age >=18.
2. Symptomatic patient: Transient ischemic attack (TIA), amaurosis fugax, or minor/non-disabling stroke (in the hemisphere supplied by the target vessel) within 180 days of enrollment; asymptomatic patient: meets angiographic and clinical inclusion criteria.
3. Patient has no childbearing potential or a negative pregnancy test within 30 days of study procedure.
4. Patient or legally authorized representative, and the patient's physician, agree to have the patient return for all required clinical contacts following study enrollment.
5. Patient or legally authorized representative has been informed of the nature of the study, and has provided written informed consent, approved by the appropriate Institutional Review Board (IRB)/Medical Ethics Committee (MEC) of the respective clinical site. (Sample consent - Appendix A-2).
6. Patient must meet two or more of the criteria listed in a-e OR one or more of the criteria listed in f-q below:

   1. Knowledge of two or more proximal or major diseased coronary arteries with >=70% stenosis that have not, or cannot be revascularized;
   2. Unstable angina defined as rest angina with ECG changes;
   3. MI within the previous 30 days and current need for carotid artery revascularization
   4. Concurrent requirement for aortocoronary bypass or cardiac valve surgery within 30 days;
   5. Contralateral occlusion of the ICA;
   6. Currently on a list for major organ transplantation (i.e. heart, lung, liver, kidney) or is being evaluated for such;
   7. Ejection fraction <30% or New York Heart Association (NYHA) Functional Class III or higher;
   8. FEV1 <30% (Predicted);
   9. Dialysis-dependent renal failure;
   10. Uncontrolled diabetes defined as fasting glucose >400 mg/dl and ketones >2+;
   11. Restenosis after previous CEA (defined as >=50% by angiography for symptomatic patients or >=80% by angiography for asymptomatic patients);
   12. Patient is status/post radiation treatment to the neck;
   13. Patient is status/post radical neck surgery;
   14. Surgically inaccessible lesions (e.g. lesions above the level of C2 or below the clavicle, lesions obstructed by tumors in the neck);
   15. Spinal immobility - inability to flex neck beyond neutral or kyphotic deformity;
   16. Presence of tracheostomy stoma;
   17. Contralateral laryngeal nerve paralysis. Anatomic Inclusion Criteria NOTE: Angiographic measurements must be made utilizing either on-line quantitative carotid angiography (QCA) or electronic calipers with magnification correction.

1. Patient has a discrete lesion located in the ICA (with or without involvement of the contiguous CCA).

2. Carotid stenosis must be >= 50% by angiography (symptomatic patient) or >= 80% by angiography (asymptomatic patient).

3. Target ICA vessel reference diameter must be >=4.0 mm and =<9.0 mm by angiography.

NOTE: Patients with bilateral carotid stenosis are eligible. Management of the non-study stenosis may be done in accordance with local Principal Investigator recommendation. Treatment of the non-study artery must take place either >30 days before or >30 days after the study procedure is completed.

Specific for the ACCUNET System 4. Expected ability to deliver the ACCUNET System distal to the lesion (absence of excessive tortuosity) and an available straight or mildly angulated segment >= 4 cm, by angiography, in the distal ICA (prior to the petrous portion of the vessel) in which to place the embolic protection device.

5. The diameter of the straight or mildly angulated segment, in the distal ICA prior to the petrous portion of the vessel, must be >= 3.25 mm and =< 7.5 mm by angiography.

Exclusion Criteria:

Candidates will be ineligible for enrollment in the study if any one of the following conditions apply:

1. Patient has an evolving stroke.
2. Patient has history of intolerance or allergic reaction to any of the study medications or materials, including heparin, aspirin, baby aspirin, nitinol, or x-ray contrast.
3. Patient has history of intolerance or allergic reaction to both ticlopidine and clopidogrel.
4. Patient has active bleeding diathesis or coagulopathy or will refuse blood transfusions.
5. Patient has a history of major ipsilateral stroke likely to confound study endpoints.
6. Patient has severe dementia.
7. Patient has a history of spontaneous intracranial hemorrhage within the past 12 months.
8. Patient has had a recent (<7 days) stroke of sufficient size (on CT or MRI) to place him or her at risk of hemorrhagic conversion during the procedure.
9. Patient had hemorrhagic transformation of an ischemic stroke within the past 60 days.
10. Patient has Hgb < 8 gm/dl (unless on dialysis), platelet count < 50,000, uncorrected INR > 1.5, or heparin-associated thrombocytopenia.
11. Patient has any condition that precludes proper angiographic assessment or makes percutaneous arterial access unsafe (e.g. morbid obesity, sustained SBP > 180 mm Hg.).
12. Patient has had neurologic illness within the past two years characterized by fleeting or fixed neurologic deficit which cannot be distinguished from TIA or stroke (e.g. partial or secondarily generalized seizures; complicated or classic migraine; tumor or other space-occupying brain lesions; subdural hematoma, cerebral contusion or other post-traumatic lesions; intracranial infection; demyelinating disease; moderate to severe dementia; or intracranial hemorrhage).
13. Patient is actively participating in another drug or device trial (IND or IDE) that has not completed the required protocol follow-up period. Patients may be enrolled only once in the ARCHeR clinical trial and may not participate in any other clinical trial during the ARCHeR follow-up period.
14. Patient or patient's legally authorized representative is unable to understand and cooperate with study procedures or provide informed consent.
15. Patient has a life expectancy less than two years.
16. Patient has vertebrobasilar insufficiency symptoms only, without clearly identifiable symptoms referable to the targeted carotid artery
17. Knowledge of cardiac sources of emboli (e.g. left ventricular aneurysm, atrial fibrillation, intracardiac filling defect, cardiomyopathy, aortic or mitral prosthetic heart valve, cardioversion of atrial fibrillation within 30 days prior to intervention, calcific aortic stenosis, endocarditis, mitral stenosis, atrial septal defect (ASD), atrial septal aneurysm, or left atrial myxoma).
18. Patient has had a recent GI bleed that would interfere with antiplatelet therapy.

Anatomic Exclusions

1. Severe vascular tortuosity or anatomy that would preclude the safe introduction of a guide catheter, guide sheath, embolic protection system, or stent system.
2. Presence of previously placed intravascular stent or intravascular graft in the ipsilateral distribution. (Patch grafts are not an exclusion criterion.)
3. Presence of extensive or diffuse atherosclerotic disease involving the aortic arch and proximal common carotid artery that would preclude the safe introduction of a guide catheter or guide sheath.
4. An intraluminal filling defect (defined as an endoluminal lucency surrounded by contrast, seen in multiple angiographic projections, in the absence of angiographic evidence of calcification) that is not associated with an ulcerated target lesion
5. Other abnormal angiographic findings such as: ipsilateral intracranial or extracranial arterial stenosis greater in severity than the lesion to be treated, cerebral aneurysm >= 5 mm, AVM (arteriovenous malformation) of the cerebral vasculature, AV fistula, or other confounding intracranial lesion.
6. Bilateral carotid stenosis if the intervention is planned within the 30-day ARCHeR periprocedure period.
7. Occlusion [Thrombolysis In Myocardial Infarction Trial (TIMI 0)] or "string sign" >1 cm of the ipsilateral common or internal carotid artery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 581
Dates: Start 2000-05; Primary Completion 2003-10 (Actual); Study Completion 2003-11 (Actual)

PRIMARY OUTCOMES:
All Stroke, death and MI | within 30 days

SECONDARY OUTCOMES:
Ipsilateral stroke | between 31 days and 12 months
2. Target vessel revascularization | six and 12 months
3. Ultrasound evaluation | six and 12 months
4. Acute device success for the RX ACCULINK System | Acute
5. Acute device success for the RX ACCUNET Embolic Protection System | Acute
6. Clinical Success | Acute
7. Access site complications requiring treatment. | Acute

CONTACTS AND LOCATIONS:
Overall Officials: L. Nelson Hopkins, M.D., Principal Investigator — Millard Fillmore Hospital, Buffalo, NY; Mark H. Wholey, MD, Principal Investigator — Shadyside Medical Center, Pittsburgh, PA

REFERENCES:
- [Background] Naylor AR. Regarding "Protected carotid stenting in high-surgical-risk patients: the ARCHeR results". J Vasc Surg. 2007 Jan;45(1):222-3; author reply 223-4. doi: 10.1016/j.jvs.2006.08.089. No abstract available. PMID 17210414
- [Background] Gray WA, Hopkins LN, Yadav S, Davis T, Wholey M, Atkinson R, Cremonesi A, Fairman R, Walker G, Verta P, Popma J, Virmani R, Cohen DJ; ARCHeR Trial Collaborators. Protected carotid stenting in high-surgical-risk patients: the ARCHeR results. J Vasc Surg. 2006 Aug;44(2):258-68. doi: 10.1016/j.jvs.2006.03.044. PMID 16890850
- [Background] Schonholz CJ, Uflacker R, Parodi JC, Hannegan C, Selby B. Is there evidence that cerebral protection is beneficial? Clinical data. J Cardiovasc Surg (Torino). 2006 Apr;47(2):137-41. PMID 16572087
- [Background] Kasirajan K. What is the latest in inventory for carotid stenting and cerebral protection? Perspect Vasc Surg Endovasc Ther. 2005 Jun;17(2):135-41. doi: 10.1177/153100350501700217. PMID 16110380
- [Background] Gray WA. Endovascular treatment of extra-cranial carotid artery bifurcation disease. Minerva Cardioangiol. 2005 Feb;53(1):69-77. PMID 15788981
- [Background] Gray WA. A cardiologist in the carotids. J Am Coll Cardiol. 2004 May 5;43(9):1602-5. doi: 10.1016/j.jacc.2003.11.051. PMID 15120818
- [Background] Illig KA, Zhang R, Tanski W, Benesch C, Sternbach Y, Green RM. Is the rationale for carotid angioplasty and stenting in patients excluded from NASCET/ACAS or eligible for ARCHeR justified? J Vasc Surg. 2003 Mar;37(3):575-81. doi: 10.1067/mva.2003.79. PMID 12618695